CLINICAL TRIAL: NCT06601270
Title: A Registry of Spontaneous Coronary Artery Dissection
Brief Title: SCAD : a Registry of Spontaneous Coronary Artery Dissection
Acronym: SCAD
Status: Recruiting | Type: Observational
Sponsor: European Society of Cardiology (Network)
Responsible Party: Sponsor
Other Study IDs: SCAD registry
Record Dates: First submitted 2020-10-15; First posted 2024-09-19 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Spontaneous Coronary Artery Dissection
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective: There are no interventions as the study is purely observational.
  Interventions: Other: There are no interventions as the study is purely observational.
- Prospective: There are no interventions as the study is purely observational.
  Interventions: Other: There are no interventions as the study is purely observational.

INTERVENTIONS:
Other: There are no interventions as the study is purely observational. — There are no interventions as the study is purely observational.

SUMMARY:
Spontaneous coronary artery dissection (SCAD) is an increasingly recognised cause of non-atherosclerotic acute coronary syndromes (ACS), predominantly afflicting young women without conventional atherosclerotic risk factors. Knowledge of SCAD has advanced considerably in the last few years as a result of data from a number of local and national registries 1-6. Like all rarer diseases however, a better understanding of SCAD will require international collaboration. At present, there is no European or International SCAD registry despite increasing recognition that there are key differences in the diagnosis, interventional and medical management of SCAD compared with conventional atherosclerotic ACS. The ESC-ACCA Study Group on Spontaneous Coronary Artery Dissection supported by the European Observational Research Programme will now build the first pan-European SCAD registry to advance our understanding of current management of this condition, inform guidelines, educate clinical colleagues and advance research.

DETAILED DESCRIPTION:
Observational, multicentre, international retrospective and prospective cohort study.

Since this is an observational study, a formal sample size is not necessary. At least 500 prospectively recruited patients and 500 historical cases will be enrolled.

Patient data will be collected at the following time-points:

* First SCAD event visit (retrospectively on chart review)
* First follow-up: at time of enrolment
* Yearly follow-up: up to 1, 2, 3, 4 and 5 years post enrolment or until study completion

Approximately 30 countries and 120 sites will participate in this registry.

ELIGIBILITY:
Inclusion Criteria:

* Patient having signed an Informed Consent
* Patient aged 18 years and over
* SCAD clinical diagnosis within the past 10 years and available coronary angiographic imagery

Exclusion Criteria:

* Patient unwilling or unable to consent
* Patients with iatrogenic or atherosclerotic coronary dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged 18 years and over with SCAD clinical diagnosis within the past 10 years and available coronary angiographic imagery.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Patient Status: | Up to 5 years post-enrollment
  * Measure: Functional health status and clinical condition during follow-up.
  * Unit of Measure: Categorized as stable, improved, or worsened.
Vital Signs: | Up to 5 years post-enrollment
  -Heart Rate: Measure: Heart rate monitoring. Unit of Measure: Beats per minute (bpm).
  -Blood Pressure: Measure: Systolic and diastolic blood pressure measurement. Unit of Measure: Millimeters of mercury (mmHg).
  -Oxygen Saturation: Measure: Oxygen saturation monitoring. Unit of Measure: Percentage (%).
Recurrent SCAD Events: | Up to 5 years post-enrollment
  * Measure: Documentation of recurrent SCAD events, including clinical presentation, diagnosis, management, and procedures.
  * Unit of Measure: Number of recurrent SCAD events.
Imagery: | Up to 5 years post-enrollment
  * Measure: Coronary angiography anonymized and sent for central review (Corelab) for confirmation and analysis.
  * Unit of Measure: Yes/No (whether imagery was obtained and sent).
Medications: | Up to 5 years post-enrollment
  Antiplatelet Medications:
  * Measure: Use of antiplatelet medications during follow-up. Unit of Measure: Number of antiplatelet medications prescribed.
  * Beta-Blockers:
  Measure: Use of beta-blocker medications during follow-up. Unit of Measure: Number of beta-blockers prescribed.
  -ACE Inhibitors/ARBs: Measure: Use of ACE inhibitors or angiotensin receptor blockers (ARBs) during follow-up.
  Unit of Measure: Number of ACE inhibitors/ARBs prescribed.
  -Calcium Channel Blockers: Measure: Use of calcium channel blockers during follow-up. Unit of Measure: Number of calcium channel blockers prescribed.
  -Statins: Measure: Use of statin medications during follow-up. Unit of Measure: Number of statins prescribed.
  -Other Medications (if applicable): Measure: Use of other medication classes during follow-up. Unit of Measure: Number and type of additional medications prescribed.
Menstrual, Contraceptive, and Obstetric History: | Up to 5 years post-enrollment
  * Measure: Menstrual status, use of contraceptives, and obstetric history during follow-up.
  * Unit of Measure: Categorical variables (e.g., premenopausal, postmenopausal; use of contraceptives: Yes/No).
Discharge Information: | Up to 5 years post-enrollment
  * Measure: Discharge status following SCAD-related hospital admissions.
  * Unit of Measure: Categorical variables (e.g., discharged to home, transferred to rehabilitation).

SECONDARY OUTCOMES:
Procedures: | Up to 5 years post-enrollment
  * Measure: Documentation of any medical or surgical procedures related to SCAD during follow-up (e.g., coronary interventions).
  * Unit of Measure: Number of procedures.
Other Coronary Vascular Events: | Up to 5 years post-enrollment
  * Measure: Occurrence of any other coronary vascular events (e.g., myocardial infarction, ischemia, revascularization).
  * Unit of Measure: Number of events.
Symptomatology: | Up to 5 years post-enrollment
  * Measure: Patient-reported symptoms related to cardiovascular health (e.g., chest pain, dyspnea, palpitations).
  * Unit of Measure: Symptom frequency and severity (scale-based or categorical, e.g., mild, moderate, severe).
Pregnancy and Hormonal Therapy (when applicable): | Up to 5 years post-enrollment
  * Measure: Pregnancy status and use of hormonal therapy during follow-up.
  * Unit of Measure: Categorical variables (e.g., pregnant: Yes/No; hormonal therapy: Yes/No).
Exercise History: | Up to 5 years post-enrollment
  -Exercise Frequency: Measure: Frequency of exercise sessions per week. Unit of Measure: Times per week.
  -Exercise Duration: Measure: Duration of each exercise session. Unit of Measure: Minutes per session.
  -Type of Exercise: Measure: Type of physical activity performed (e.g., aerobic, resistance, flexibility).
  Unit of Measure: Categorical variables (e.g., aerobic, resistance, flexibility).
Mental Health and Wellbeing: | Up to 5 years post-enrollment
  -Anxiety (HADS-A): Measure: Anxiety levels assessed using the Hospital Anxiety and Depression Scale-Anxiety subscale (HADS-A).
  Unit of Measure: HADS-A score (range: 0 to 21; higher scores indicate worse anxiety symptoms).
  -Depression (PHQ-9): Measure: Depression levels assessed using the Patient Health Questionnaire-9 (PHQ-9).
  Unit of Measure: PHQ-9 score (range: 0 to 27; higher scores indicate worse depression symptoms).
  -Overall Wellbeing: Measure: Overall wellbeing rating on a self-reported scale. Unit of Measure: Wellbeing rating score (range: 1 to 10; higher scores indicate better wellbeing).
Employment Post-SCAD: | At first follow-up visit only
  * Measure: Employment status following SCAD event.
  * Unit of Measure: Categorical variables (e.g., employed, unemployed, part-time).

CONTACTS AND LOCATIONS:
Overall Officials: Adham GHARIEB, PharmD, Study Director — ESC
Locations (73):
- ICBA - Instituto Cardiovascular de Buenos Aires, Buenos Aires, Argentina
- Austria (5):
  - Medical University of Innsbruck, Internal Medicine III, Innsbruck
  - Klinik Landstrasse, Vienna
  - Klinik Ottakring, Vienna
  - Medical University of Vienna, Vienna
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Belgium (12):
  - AZ Sint jan, current president of Belgian ACCA, Bruges
  - Cliniques Universitaires Saint-Luc (UCL), Brussels
  - Universitair Ziekenhuis Brussels, Brussels
  - Antwerp University Hospital, Edegem
  - Ziekenhuis Oost Limburg, Interventional cardiology/Coronary Care, Genk
  - AZ Sint Lucas hospital, Ghent
  - Ghent University Hospital, Ghent
  - University Hospitals Leuven, Leuven
  - CHR La Citadelle, Liège
  - Les cliniques Saint Pierre, Ottignies
  - AZ Delta, Roeselare
  - AZ Nikolaas, Sint-Niklaas
- Clinical Center University of Sarajevo, Sarajevo, Bosnia and Herzegovina
- Brazil (3):
  - Hospital Israelita Albert Einstein, São Paulo
  - Instituto do Coração do HCFMUSP, São Paulo
  - Universidade Federal de São Paulo (UNIFESP), São Paulo
- University Hospital of Split (KBC Split), Split, Croatia
- Nicosia General Hospital, Nicosia, Cyprus
- Czechia (2):
  - Nemocnice Pardubického kraje, Pardubice
  - Hospital Na Homolce, Prague
- Denmark (4):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Hellerup
  - Odense University Hospital, Odense
- France (6):
  - CHRU Jean Minjoz, Besançon
  - Gabriel Montpied Hospital - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital de Chartres Louis Pasteur, Le Coudray
  - Cardiovascular Hospital Louis Pradel - Hospices Civils de Lyon, Lyon
  - Hôpital Jacques Cartier, Massy
  - Hôpital Cardiologique du Haut Lévêque - Bordeaux University, Pessac
- Germany (4):
  - Schüchtermann-Klinik Bad Rothenfelde, Bad Rothenfelde
  - Vivantes Klinikum in Friedrichshain, Berlin
  - University Heart and Vascular Center Hamburg Eppendorf, Hamburg
  - Robert Bosch Hospital, Stuttgart
- Greece (2):
  - Sotiria Thoracic Diseases Hospital, Athens
  - General Hospital of Kozani, Kozani
- Tehran Heart Center, Tehran, Iran
- Italy (8):
  - Papa Giovanni XXIII Azienda Ospedaliera, Bergamo
  - Policlinico Riuniti Foggia, Foggia
  - Ospedale Policlinico San Martino IRCCS, Genova & Università di Genova, Genoa
  - Presidio Ospedaliero Carlo Poma, Mantova
  - ASST Grande Ospedale Niguarda, Milan
  - Centro Cardiologico Monzino, IRCCS, Milan
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
- Netherlands (3):
  - Noordwest Ziekenhuisgroep / NorthWest Clinics, Alkmaar
  - Amphia Hospital, Breda
  - Radboud University Medical Centre, Nijmegen
- Auckland City Hospital - Green Lane Cardiovascular Service, Auckland, New Zealand
- Haukeland University Hospital - Invasive cardiology, Bergen, Norway
- Institute of Cardiology - Department of Interventional Cardiology and Angiology, Warsaw, Poland
- Portugal (4):
  - Hospital Fernando Fonseca, Amadora
  - Hospital de Braga, Braga
  - Hospital do Espirito Santo de Evora, Evora
  - Centro Hospitalar Tondela Viseu, Tondela
- Serbia (2):
  - University Hospital Centre Bezanijska Kosa, Belgrade
  - Cardiology Clinic, UCC Nis, Niš
- National University Heart Centre Singapore, Singapore, Singapore
- Stredoslovensky ustav srdcovych a cievnych chorob a.s, Banská Bystrica, Slovakia
- Hospital Universitario de la Princesa, Madrid, Spain
- United Kingdom (7):
  - William Harvey Hospital, Ashford
  - Glan Clwyd Hospital, Bodelwyddan
  - Bournemouth Hospital, Bournemouth
  - Bristol Heart Institute, Bristol
  - University Hospitals, Leicester
  - Royal Brompton & Chelsea & Westminster Hospital, London
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No